CLINICAL TRIAL: NCT04056936
Title: The Scope of Tongue-tie in Norway: Its Prevalence and Consequences for Child Health
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Oslo (Other)
Collaborators: The Hospital of Vestfold (Other); Oslo University Hospital (Other); Sykehuset Telemark (Other Government)
Responsible Party: Principal Investigator, Atle Klovning, MD. PhD. Associate Professor, University of Oslo
Other Study IDs: 2018/FO201556
Record Dates: First submitted 2019-06-24; First posted 2019-08-14 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Tongue Tie; Ankyloglossia
Keywords: Breastfeeding; Lactational mastitis; Infant nutrition; Infant growth; Speech development; Frenotomy
MeSH Terms: conditions — Ankyloglossia; Breast Feeding | interventions — Oral Frenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infants diagnosed with a tongue-tie and a frenotomy: If a tongue-tie is present at the routine newborn examination, the infant can be included in the study. If the infant also has breastfeeding problems and there is a decreased tongue mobility and poor sucking ability, the pediatrician may find indication for frenotomy. If the frenotomy is performed before discharge the infant is included in this group. All Mother-infant dyads will get breastfeeding support.
  Interventions: Procedure: Frenotomy
- Infants diagnosed with a tongue-tie and no frenotomy: The infants that are recruited to the tongue-tie cohort that do not receive treatment before discharge. The pediatrician evaluates that the tongue tie does not cause any functional problems and no treatment is performed before discharge. All Mother-infant dyads will get breastfeeding support.
- All infants born in Telemark and Vestfold Counties: All the infants born in the study period that will contribute to the prevalence study.

INTERVENTIONS:
Procedure: Frenotomy — To map the severity determining any possible consequences a tongue-tie may have for breastfeeding and infant nutrition we will follow-up a cohort of tongue-tied infants to register if the feeding, growth, thriving and speech of the infant/child is affected by a tongue-tie.
  Other Names: Breastfeeding support
  Groups: Infants diagnosed with a tongue-tie and a frenotomy

SUMMARY:
The study is a prospective multi-centre clinical follow-up study of prevalence and severity of tongue-tie in neonates in Norway. During one year around 2600 newborn infants will be examined for tongue-tie in the two participating hospitals. The infants diagnosed with a tongue tie, will be followed to assess the proportion of infants treated and the severity. Feeding outcomes will be observed up to 6 months of age.

DETAILED DESCRIPTION:
A tongue-tie may cause problems for child and mother. There are no previous studies from Norway that have assessed the magnitude and severity of tongue-tie in infants. The prevalence of tongue-tie in Norway and to what degree it influences mother and child health is unknown. It is of great importance to address a problem with possible negative effect on breastfeeding and maternal and child health. Current clinical practice varies due to incomplete knowledge of the condition. An unknown proportion of infants with tongue-tie may not be diagnosed or receive treatment. Current international research recommends treatment of tongue-tie if it causes breastfeeding problems. This project will add significant knowledge about tongue-tie in Norway.

The project supports:

* Filling knowledge gaps by researching the prevalence and severity of the condition.
* Obtaining new knowledge for the health services by establishing assessment of tongue-tie prevalence in Norway. This can be used for planning of the healthcare services.
* Improving existing practice by describing the condition and implementing best practice diagnosis and treatment.
* Creating societal benefits by improving infant nutrition and maternal health.

During the year of the study, the pediatricians at each hospital will assess the prevalence of tongue-tie in all newborn infants in their hospital. The examination will be part of the standard newborn examination which usually takes place during the 2nd day of life. A simple and short registration form will be filled out electronically, noting the type of tongue-tie and symptoms for each infant with the diagnosis. In addition, the diagnosis Ankyloglossia Q38.1 will be registered in the electronic journal system. The examination of the infant's mouth is completely safe and is already performed to asses if there is a cleft palate. The pediatrician will examine the area under the tongue in addition to the palate. All newborn infants will be examined to obtain a trustworthy prevalence. If a frenotomy is required and performed, this will be registered in the registration form and the procedure code for frenotomy EJC 20 will be registered in the electronic journal system. The breastfeeding self-efficacy tool (BSES-SF) is used for patient reported outcome measures.as well as WHO's breastfeeding indicators

To map the severity determining any possible consequences a tongue-tie may have for breastfeeding and infant nutrition the investigators will follow-up a cohort of tongue-tied infants to register if the feeding, growth, thriving and speech of the infant/child is affected by a tongue-tie.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be born in a participating hospital during the study period.
* Subjects that are recruited for follow-up must have a diagnose of tongue-tie as determined by the pediatrician in the hospital.
* Infants with a tongue-tie that have been treated with a frenotomy and infants that have not received treatment.

Exclusion Criteria:

* Infants where the parents do not wish to participate in the study or where the parents do not to understand English or Norwegian.

Ages: 1 Day to 2 Weeks | Sex: All
Age Groups: Child
Study Population: Infants 0 days to 2 weeks old diagnosed with a tongue tie in the counties of Telemark and Vestfold during the study enrollment period September 2019 - August 2020.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ankyloglossia in Norway | September 2019 - August 2021
  The to assess the prevalence of tongue-tie in newborn infants in Norway.

SECONDARY OUTCOMES:
Proportion of infants treated with a frenotomy | September 2019 - December 2021
  The number of infants treated on indication after the standardized diagnostic approach and the method of treatment have been introduced in the centers of intervention.
Variations in diagnosis of tongue tie and breastfeeding outcomes | September 2019 - December 2021
  Number of infants with the diagnosis Q38.1 in the intervention counties compared to counties that are not a part of the study.
Severity of breastfeeding problems | September 2019 - December 2021
  Breastfeeding problems and the duration of exclusive breastfeeding measured in months in the tongue tied infants that receive treatment compared to those who are not treated.
Adverse events | September 2019 - December 2021
  Severity of adverse events related to the treatment of the infant as assessed by CTCAE v5.0.

OTHER OUTCOMES:
Long term followup - Breastfeeding duration and introduction of solids | September 2019 - August 2023
  Duration of any breastfeeding in months and any problems with the introduction of solids is mapped 3 years after inclusion in the study.
Long term followup - Speech development | September 2019 - August 2023
  Problems with child's speech development at the age of 3 years. Referral to treatment by Speech Language Pathologist.

CONTACTS AND LOCATIONS:
Overall Officials: Atle Klovning, MD. PhD, Study Director — University of Oslo

IPD SHARING:
Plan to Share IPD: No